CLINICAL TRIAL: NCT04663256
Title: Effectiveness of a Cognitive Stimulation Program on Anxiety, Depression and Quality of Life in People Older Than 70 Years With Mild Cognitive Impairment.
Brief Title: Effects of Cognitive Stimulation in Older People With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén_2020
Record Dates: First submitted 2020-11-15; First posted 2020-12-10 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Mild Cognitive Impairment; Older People
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Stimulation Group (Experimental): This group receives physical training based on exercises for cognitive stimulation.
  Interventions: Other: Cognitive stimulation group
- Control Group (No Intervention): This group does not receive any treatment.

INTERVENTIONS:
Other: Cognitive stimulation group — Each week for 12 weeks, GE participants attend three 60-minute sessions of cognitive exercises.
  Arms: Cognitive Stimulation Group

SUMMARY:
Mild cognitive impairment is becoming one of the most common cynical manifestations that affect older people. That is why there is a need to investigate non-pharmacological interventions that help to improve or maintain this problem.

DETAILED DESCRIPTION:
Each week for 12 weeks, GE participants will attend three 60-minute sessions of cognitive exercises. Each session is divided into 10 minutes of memory practice, which includes short-term and long-term memory; 10 minutes of language skills, including vocabulary, comprehension, reading and writing exercises; 10 minutes of calculation, in which arithmetic, similar and different operations are carried out; 10 minutes of praxis and gnosis where drawing and recognition and auditory, tactile, spatial, visual attention were promoted; 10 minutes of orientation where knowledge of space, person and place is developed; and 10 minutes of executive functions in which exercises of organization, planning and problem solving are worked.

ELIGIBILITY:
Inclusion Criteria:

* With or without dependency to move.
* People who show mild cognitive impairment.
* That they were able to carry out the different selected questionnaires.

Exclusion Criteria:

* People with visual deficit.
* People already enrolled in a cognitive program.
* Score between 24 and 10 in the Mini Cognitive Exam (MEC).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
MMSE (mini-mental state examination) | Baseline-8 weeks
  A tool that can be used to systematically and thoroughly assess mental status.
Yesavage Geriatric Depression Scale Adjetivo 1 relating to old people, especially with regard to their healthcare. a geriatric hospital Sustantivo 1 an old person, especially one receiving special care. a rest home for geriatrics. | Baseline-8 weeks
  Hetero-administered questionnaire used to detect depression in people over 65 years of age.
Hamilton Scale for Anxiety. | Baseline-8 weeks
  Hetero-administered scale used for the detection of anxiety, exploring the interruption of the emotional continum and subjective feelings of tension, restlessness or nervousness.
SF-36 (The Short Form-36 Health Survey) | Baseline-8 weeks
  Used extensively for assessing health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- U.E.D. Virgen de la Capilla, Jaén, Spain